CLINICAL TRIAL: NCT04547972
Title: The Effects of Higher- And Lower-Load Resistance Exercise Training on Leg and Arm Skeletal Muscle Mass in Healthy Young Adult Females
Brief Title: The Effects of Heavier- and Lighter-load Resistance Training on Arm and Leg Muscle Mass in Young Adult Women
Acronym: FHALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Cameron Mitchell, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H20-01570
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Skeletal Muscle Hypertrophy
Keywords: Skeletal Muscle; Hypertrophy; Strength; Muscle Endurance
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Intervention Model Description: A within participant design will be used wherein each participant will be assigned to both training conditions. One arm and one leg will train with higher-loads and one arm and one leg will train with lower-loads; limb allocation will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher-load limbs (Active Comparator): This treatment arm will have participants performing resistance training with loads of ~80% of an individuals one-repetition maximum. Each participant will have one arm and one leg assigned to this condition.
  Interventions: Other: Higher-load resistance training
- Lower-load limbs (Active Comparator): This treatment arm will have participants performing resistance training with loads of ~30% of an individuals one-repetition maximum. Each participant will have one arm and one leg assigned to this condition.
  Interventions: Other: Lower-load resistance training

INTERVENTIONS:
Other: Higher-load resistance training — This intervention will have one arm and one leg of each participant training with ~80% of their one repetition maximum
  Arms: Higher-load limbs
Other: Lower-load resistance training — This intervention will have one arm and one leg of each participant training with ~30% of their one repetition maximum
  Arms: Lower-load limbs

SUMMARY:
When you perform weightlifting, your body makes new proteins within your muscle. These new proteins can increase the size of the fibers within your muscle to make your muscle larger, a process called hypertrophy. The common convention surrounding gains in muscle mass and strength are that higher-loads (i.e. heavier weights) used for fewer repetitions are better for increasing strength and lower-loads (i.e. lighter weights) used for higher repetitions are better for increasing muscle mass. However, recent research has found that when higher- and lower-loads are used when participants exercise until volitional fatigue (i.e. cannot perform another repetition), muscle mass and strength increases are similar regardless of using a higher- or lower-load. Many of these studies have examined this effect in males with fewer studies examining the effects of higher- and lower-load training in females when assessing changes in muscle mass, strength, and muscle endurance.

Further, it has been shown that there is substantial individual variation in response to resistance exercise training where individuals can be broadly categorized as higher- or lower-responders to resistance exercise training. This study aims to explore how the muscle mass, strength, and muscle endurance of females are impacted by both higher- and lower-loads while also exploring how individuals may respond to the training interventions.

DETAILED DESCRIPTION:
The study will be a total of 12 weeks in total duration. Weeks 1 and 12 will include testing assessments of skeletal muscle mass, muscle strength, and muscle endurance. Weeks 2-11 will be comprised of the resistance training intervention wherein participants will train thrice weekly at the Chan Gunn Pavilion research laboratory at the University of British Columbia.

Resistance training sessions will include unilateral knee extensions and unilateral dumbbell bicep preacher curls with each being performed for three sets. Limbs assigned to train with higher-loads will perform between 8-12 repetitions per set and limbs assigned to train with lower-loads will perform between 20-25 repetitions per set. Participants will rest 90 seconds between sets and 120 seconds between exercises. Each exercise will be performed in its entirety before moving on to the next.

Participants will also be supplemented with whey protein which will be ingested twice daily during the resistance training phase.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 18-30 years of age
3. Can fluently read and write in English
4. Able to commit to three training sessions per week for a continuous 10-week period as well as testing one week before and one week after this 10-week training period
5. All "No" answers on the Canadian Society for Exercise Physiology Get Active questionnaire or doctors' approval to participate

Exclusion Criteria:

1. Allergic to dairy products or are lactose-intolerant (participants will be supplemented with whey protein twice daily for the 10-week training period)
2. Allergic to any of the following ingredients which are present in the whey protein concentrate supplement: Bos taurus - Milk, Cocoa, Natural and Artificial Flavours, Xanthan Gum, Sucralose, Non-genetically modified organism Sunflower Lecithin
3. Any major uncontrolled cardiovascular, muscular, metabolic, and/or neurological disorders
4. Lung or kidney disease
5. Medical conditions impacting on their ability to undertake strenuous physical activity
6. Regular use of any mental health medications that may lead to excessive weight gain (selective serotonin reuptake inhibitors, second generation antipsychotics, antiepileptic drugs)
7. Participated in consistent resistance exercise training more than twice per month in the previous 12 months
8. Participated in consistent vigorous aerobic training more than twice per week in the previous 12 months
9. Significant gain or loss of body mass in the past 6 months (greater than 2 kg)
10. Current smoker
11. BMI less than 18 or over 30

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Change in upper- and lower-body skeletal muscle mass between weeks 1 and 12 | Weeks 1 and 12
  The total skeletal muscle mass measured in each individual arm and leg quantified using dual-energy x-ray absorptiometry scanning

SECONDARY OUTCOMES:
Change in unilateral dumbbell bicep preacher curl one repetition maximum between weeks 1 and 12 | Weeks 1 and 12
  The maximum amount of weight that an individual can move for one full repetition during the unilateral dumbbell bicep preacher curl exercise
Change in unilateral knee extension one repetition maximum between weeks 1 and 12 | Weeks 1 and 12
  The maximum amount of weight that an individual can move for one full repetition during the unilateral knee extension exercise
Change in unilateral dumbbell bicep preacher curl relative muscle endurance between weeks 1 and 12 | Weeks 1 and 12
  The maximum number of repetitions that can be completed with 30% and 80% of the individuals current one repetition maximum for the unilateral dumbbell bicep preacher curl exercise
Change in unilateral dumbbell bicep preacher curl absolute muscle endurance between weeks 1 and 12 | Weeks 1 and 12
  The maximum number of repetitions that can be completed with 30% and 80% of the individuals baseline one repetition maximum for the unilateral dumbbell bicep preacher curl exercise
Change in unilateral knee extension relative muscle endurance between weeks 1 and 12 | Weeks 1 and 12
  The maximum number of repetitions that can be completed with 30% and 80% of the individuals current one repetition maximum for the unilateral knee extension exercise
Change in unilateral knee extension absolute muscle endurance between weeks 1 and 12 | Weeks 1 and 12
  The maximum number of repetitions that can be completed with 30% and 80% of the individuals baseline one repetition maximum for the unilateral knee extension exercise
Change in Vastus Lateralis and Biceps Brachii Cross Sectional Area between weeks 1 and 12 | Weeks 1 and 12
  The cross sectional area of the vastus lateralis and biceps brachii muscles measured using ultrasonography
Change in Vastus Lateralis and Biceps Brachii Muscle Thickness between weeks 1 and 12 | Weeks 1 and 12
  The thickness of the vastus lateralis and biceps brachii muscles measured using ultrasonography
Change in Vastus Lateralis Pennation Angle between weeks 1 and 12 | Weeks 1 and 12
  The pennation angle of the vastus lateralis muscle fibers measured using ultrasonography
Change in Vastus Lateralis Fascicle Length between weeks 1 and 12 | Weeks 1 and 12
  The length of the fascicles of the vastus lateralis muscle measured using ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Cameron J Mitchell, PhD, Principal Investigator — University of British Columbia
Locations (1):
- The University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
A plan has not yet been made to make individual participant data available to other researchers

REFERENCES:
- [Background] Campos GE, Luecke TJ, Wendeln HK, Toma K, Hagerman FC, Murray TF, Ragg KE, Ratamess NA, Kraemer WJ, Staron RS. Muscular adaptations in response to three different resistance-training regimens: specificity of repetition maximum training zones. Eur J Appl Physiol. 2002 Nov;88(1-2):50-60. doi: 10.1007/s00421-002-0681-6. Epub 2002 Aug 15. PMID 12436270
- [Background] Schoenfeld BJ, Grgic J, Ogborn D, Krieger JW. Strength and Hypertrophy Adaptations Between Low- vs. High-Load Resistance Training: A Systematic Review and Meta-analysis. J Strength Cond Res. 2017 Dec;31(12):3508-3523. doi: 10.1519/JSC.0000000000002200. PMID 28834797
- [Background] Mitchell CJ, Churchward-Venne TA, West DW, Burd NA, Breen L, Baker SK, Phillips SM. Resistance exercise load does not determine training-mediated hypertrophic gains in young men. J Appl Physiol (1985). 2012 Jul;113(1):71-7. doi: 10.1152/japplphysiol.00307.2012. Epub 2012 Apr 19. PMID 22518835
- [Background] Roberts BM, Nuckols G, Krieger JW. Sex Differences in Resistance Training: A Systematic Review and Meta-Analysis. J Strength Cond Res. 2020 May;34(5):1448-1460. doi: 10.1519/JSC.0000000000003521. PMID 32218059
- [Background] Franco CMC, Carneiro MADS, Alves LTH, Junior GNO, de Sousa JFR, Orsatti FL. Lower-Load is More Effective Than Higher-Load Resistance Training in Increasing Muscle Mass in Young Women. J Strength Cond Res. 2019 Jul;33 Suppl 1:S152-S158. doi: 10.1519/JSC.0000000000002970. PMID 30640303
- [Derived] Fliss MD, Stevenson J, Mardan-Dezfouli S, Li DCW, Mitchell CJ. Higher- and lower-load resistance exercise training induce load-specific local muscle endurance changes in young women: a randomised trial. Appl Physiol Nutr Metab. 2022 Dec 1;47(12):1143-1159. doi: 10.1139/apnm-2022-0263. Epub 2022 Aug 26. PMID 36027601